CLINICAL TRIAL: NCT03580369
Title: A Multi-center, Randomized, Double-blind, Active and Placebo-controlled Study to Investigate the Safety and Efficacy of Ligelizumab (QGE031) in the Treatment of Chronic Spontaneous Urticaria (CSU) in Adolescents and Adults Inadequately Controlled With H1-antihistamines
Brief Title: A Phase III Study of Safety and Efficacy of Ligelizumab in the Treatment of CSU in Adolescents and Adults Inadequately Controlled With H1-antihistamines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031C2302; 2018-000839-28 (EudraCT Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Anti-IgE; CSU; chronic spontaneous urticaria; hives severity score; itch severity score; urticaria activity score
MeSH Terms: conditions — Chronic Urticaria | interventions — ligelizumab; Omalizumab

STUDY DESIGN:
Intervention Model Description: This was a Phase III multi-center, randomized, double-blind, active- and placebo-controlled, parallel-group study. There was a screening period of up to 28 days, a 52 week double-blind treatment period, and a 12 week post-treatment follow-up period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, investigator staff and personnel performing the study assessments remained blinded to the identity of the treatment from the time of randomization until final database lock. The study drug was prepared by an independent unblinded pharmacist (or authorized delegate) and administered by an independent unblinded study drug administrator. Neither the unblinded pharmacist nor the unblinded study drug administrator was involved in any assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ligelizumab 120 mg (Experimental): Ligelizumab 120 mg arm: 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
  Interventions: Biological: Ligelizumab
- Ligelizumab 72 mg (Experimental): Ligelizumab 72 mg arm: 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
  Interventions: Biological: Ligelizumab
- Omalizumab 300 mg (Active Comparator): Omalizumab 300 mg arm: 2 injections of 1.2 mL omalizumab q4w
  Interventions: Biological: Omalizumab
- Placebo (Placebo Comparator): Placebo-ligelizumab arm: 2 injections of 1.0mL of ligelizumab placebo from Week 0 through Week 20; 1 injection of 1.0mL of ligelizumab 120 mg + 1 injection of 1.0 mL ligelizumab placebo from Week 24 through Week 48
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ligelizumab — Liquid in vial
  Arms: Ligelizumab 120 mg; Ligelizumab 72 mg
Biological: Omalizumab — Lyophilized powder for solution in vial
  Arms: Omalizumab 300 mg
Other: Placebo — Liquid in vial
  Arms: Placebo

SUMMARY:
The purpose of this study was to establish safety and efficacy of ligelizumab in adolescent and adult subjects with Chronic Spontaneous Urticaria (CSU) who remain symptomatic despite standard of care treatment by demonstrating better efficacy over omalizumab and over placebo.

The study population consisted of 1,072 male and female subjects aged ≥ 12 years who were diagnosed with CSU and who remained symptomatic despite the use of H1-antihistamines.

This was a multi-center, randomized, double-blind, active- and placebo-controlled, parallel-group study. There was a screening period of up to 28 days, a 52 week double-blind treatment period, and a 12 week post-treatment follow-up period.

DETAILED DESCRIPTION:
This was a Phase III multi-center, randomized, double-blind, active and placebo-controlled, parallel-group study. The study consisted of 3 distinct periods:

* Screening period (Day -28 to Day 1): Duration of up to 4 weeks in which subjects who have given informed consent were assessed for eligibility.
* Double-blind treatment period (52 weeks): The subjects were seen in the clinic every 4 weeks.
* Post-treatment follow-up period (12 weeks): This period consists of 3 visits (every 4 weeks) with the final visit occurring 16 weeks after the last dose at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study. The subject's, parent's or legal guardian's signed written informed consent and child's assent, if appropriate, must be obtained before any assessment is performed. Of note, if the subject reaches age of consent (age as per local law) during the study, they will also need to sign the corresponding study Informed Consent Form (ICF) at the next study visit.
* Male and female subjects ≥ 12 years of age at the time of screening.
* CSU diagnosis for ≥ 6 months.
* Diagnosis of CSU refractory to H1-AH at approved doses at the time of randomization, as defined by all of the following:
* The presence of itch and hives for ≥ 6 consecutive weeks at any time prior to Visit 1 (Day - 28 to Day -14) despite current use of non-sedating H1-antihistamine
* UAS7 score (range 0-42) ≥ 16 and HSS7 (range 0-21) ≥ 8 during the 7 days prior to randomization (Visit 110, Day 1)
* Subjects must be on H1-antihistamine at only locally label approved doses for treatment of CSU starting at Visit 1 (Day -28 to Day -14)
* Willing and able to complete a daily symptom eDiary for the duration of the study and adhere to the study visit schedules.

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or their excipients or to drugs of similar chemical classes (i.e. to murine, chimeric or human antibodies).
* Subjects having a clearly defined cause of their chronic urticaria, other than CSU. This includes, but is not limited to, the following: symptomatic dermographism (urticaria factitia), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic- or contact-urticaria.
* Diseases, other than chronic urticaria, with urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency).
* Subjects with evidence of helminthic parasitic infection as evidenced by stools being positive for a pathogenic organism according to local guidelines. All subjects will be screened at Visit 1. If stool testing is positive for pathogenic organism, the subject will not be randomized and will not be allowed to rescreen.
* Any other skin disease associated with chronic itching that might influence in the investigators opinion the study evaluations and results (e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.).
* Prior exposure to ligelizumab or omalizumab.
* H1-AH used as background medication at greater than locally label-approved doses after visit 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (141):
- United States (29):
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Greenacres City, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Clarkston, Michigan
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Pflugerville, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, South Burlington, Vermont
- Argentina (7):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Capital Federal
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Brazil (4):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Alphaville Barueri, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (7):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Zagreb, Croatia
- Czechia (4):
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Pilsen
- Denmark (2):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Herlev
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Trévenans
- Germany (12):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Szeged, Csongrád megye
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
- India (5):
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Navi Mumbai, Maharashtra
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Vijayawada
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, George Town, Pulau Pinang
- Novartis Investigative Site, Muscat, Oman
- Peru (2):
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
- Poland (6):
  - Novartis Investigative Site, Ksawerów, POL
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (6):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
- Novartis Investigative Site, Singapore, Singapore
- South Africa (3):
  - Novartis Investigative Site, Cape Town, Western Province
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
- South Korea (9):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Barcelona
- Novartis Investigative Site, Malmo, Sweden
- Thailand (3):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok, Phayathai
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Okmeydanı
  - Novartis Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Maurer M, Ensina LF, Gimenez-Arnau AM, Sussman G, Hide M, Saini S, Grattan C, Fomina D, Rigopoulos D, Berard F, Canonica GW, Rockmann H, Irani C, Szepietowski JC, Leflein J, Bernstein JA, Peter JG, Kulthanan K, Godse K, Ardusso L, Ukhanova O, Staubach P, Sinclair R, Gogate S, Thomsen SF, Tanus T, Ye YM, Burciu A, Barve A, Modi D, Scosyrev E, Hua E, Letzelter K, Varanasi V, Patekar M, Severin T; PEARL-1 and PEARL-2 trial investigators. Efficacy and safety of ligelizumab in adults and adolescents with chronic spontaneous urticaria: results of two phase 3 randomised controlled trials. Lancet. 2024 Jan 13;403(10422):147-159. doi: 10.1016/S0140-6736(23)01684-7. Epub 2023 Nov 23. PMID 38008109
- See also: A Plain Language Trial Summary is available on novctrd.com. — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,072 participants enrolled at 164 sites in 28 countries
Pre-assignment Details: There were 1,034 adult subjects and 38 adolescent subjects
Groups:
- Ligelizumab 72 mg - Adults; Ligelizumab 72 mg - Adolescents: Ligelizumab 72 mg arm: 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 120 mg - Adults; Ligelizumab 120 mg - Adolescents: Ligelizumab 120 mg arm: 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Omalizumab 300 mg - Adults; Omalizumab 300 mg - Adolescents: Omalizumab 300 mg arm: 2 injections of 1.2 mL omalizumab q4w
- Placebo - Ligelizumab 120mg - Adults: This is when patients switched to Ligelizumab: 2 injections of 1.0 mL of ligelizumab placebo q4w from Week 0 to Week 20; 1.0 mL of ligelizumab 120 mg + 1.0 mL of ligelizumab placebo q4w from Week 24 through Week 48
- Placebo - Ligelizumab 120mg - Adolesecents: 2 injections of 1.0 mL of ligelizumab placebo q4w from Week 0 to Week 20; 1.0 mL of ligelizumab 120 mg + 1.0 mL of ligelizumab placebo q4w from Week 24 through Week 48
Period: Overall Study
Arm/Group | Ligelizumab 72 mg - Adults | Ligelizumab 72 mg - Adolescents | Ligelizumab 120 mg - Adults | Ligelizumab 120 mg - Adolescents | Omalizumab 300 mg - Adults | Omalizumab 300 mg - Adolescents | Placebo - Ligelizumab 120mg - Adults | Placebo - Ligelizumab 120mg - Adolesecents
Started | 307 | 10 | 312 | 12 | 309 | 13 | 106 | 3
Completed | 263 | 10 | 258 | 9 | 267 | 10 | 91 | 3
Not Completed | 44 | 0 | 54 | 3 | 42 | 3 | 15 | 0
Not completed — No treatment due to mis-randomization | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Reason unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Technical problems | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Pregnancy | 2 | 0 | 3 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0 | 3 | 0 | 1 | 0
Not completed — Physician Decision | 4 | 0 | 4 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 7 | 0 | 2 | 0 | 3 | 0
Not completed — Protocol Violation | 6 | 0 | 6 | 1 | 8 | 2 | 1 | 0
Not completed — Adverse Event | 7 | 0 | 14 | 1 | 6 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 17 | 0 | 16 | 1 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
  Adults (1,034) + Adolescents (38) = Total (1,072)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 120 mg | Ligelizumab 72 mg | Omalizumab 300 mg | Placebo | Total
Number analyzed (Participants) | 317 | 324 | 322 | 109 | 1072
Age, Categorical [Count of Participants; unit: Participants] — Adults (971+63=1,034) + Adolescents (38) = Total (1,072) Population: Randomized Set
  Participants
    <=18 years | 10 | 12 | 13 | 3 | 38
    Between 18 and 65 years | 288 | 297 | 291 | 95 | 971
    >=65 years | 19 | 15 | 18 | 11 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
  Adults (1,034) + Adolescents (38) = Total (1,072)
  Years
    Adults: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adults | 42.3 (13.48) | 43.3 (13.12) | 42.2 (13.19) | 43.2 (14.06) | 42.7 (13.34)
    Adolescents: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescents | 14.6 (2.01) | 15.1 (1.62) | 14.7 (1.65) | 15.3 (2.08) | 14.8 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Adults (1,034) + Adolescents (38) = Total (1,072) Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to. Adults (1,034) + Adolescents (38) = Total (1,072)
  Participants
    Adult: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult: Female | 217 | 226 | 218 | 76 | 737
    Adult: Male | 90 | 86 | 91 | 30 | 297
    Adolescent: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent: Female | 5 | 9 | 9 | 1 | 24
    Adolescent: Male | 5 | 3 | 4 | 2 | 14
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to. Adults (1,034) + Adolescents (38) = Total (1,072)
  Participants
    Adult White: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult White | 226 | 220 | 221 | 80 | 747
    Adolescent White: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent White | 8 | 8 | 8 | 2 | 26
    Adult Black or African American: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Black or African American | 1 | 4 | 9 | 1 | 15
    Adolescent Black or African American: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent Black or African American | 0 | 1 | 0 | 0 | 1
    Adult Asian: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Asian | 60 | 72 | 64 | 22 | 218
    Adolescent Asian: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent Asian | 0 | 3 | 2 | 0 | 5
    Adult Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
    Adolescent Native Hawaiian or Pacific Islander: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
    Adult Native American: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Native American | 12 | 10 | 9 | 3 | 34
    Adolescents Native American: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescents Native American | 2 | 0 | 3 | 1 | 6
    Adult Multi-racial: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Multi-racial | 6 | 4 | 6 | 0 | 16
    Adolescent Multi-racial: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent Multi-racial | 0 | 0 | 0 | 0 | 0
    Adult Race Not Reported: number analyzed (Participants) | 307 | 312 | 309 | 106 | 1034
    Adult Race Not Reported | 2 | 1 | 0 | 0 | 3
    Adolescent Race Not Reported: number analyzed (Participants) | 10 | 12 | 13 | 3 | 38
    Adolescent Race Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in UAS7 at Week 12 (Multiple Imputation) of Adult Subjects
Description: The Urticaria Activity Score (UAS) is sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is sum of the HSS7 and the ISS7 scores. Possible range of weekly UAS7 score is 0 to 42. Complete UAS7 response is UAS7 = 0.
  Hives Severity Score (HSS) scale is 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. Possible range of the weekly score is therefore 0 to 21. Hives Severity Score scale: 0 - None 1 - Mild (1-6 hives/12 hours) 2 - Moderate (7-12 hives/12 hours) 3 - Severe (>12 hives/12 hours).
  Itch Severity Score (ISS) scale is 0 to 3. Score (ISS7) is derived by adding up average daily scores of 7 days preceding visit. Possible range of weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate).
  Negative change from baseline indicates improvement
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized Adult subjects who received at least one dose of study drug. Subjects were analyzed according to the treatment to which they were assigned at randomization. FAS was used for all efficacy variables, unless otherwise stated.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 306 | 312 | 306 | 106
Score | -19.368 (0.668) | -19.330 (0.660) | -20.040 (0.663) | -11.366 (1.129)
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Treatment contrast in LS mean (change), Adults; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -8.002, 95% CI 2-sided [-10.576 to -5.428], Standard Error of Mean 1.313
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Treatment contrast in LS mean (change), Adults; Test type: Superiority; p = 0.7628, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS mean = 0.672, 95% CI 2-sided [-1.169 to 2.513], Standard Error of Mean 0.939
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Treatment contrast in LS mean (change), Adults; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -7.964, 95% CI 2-sided [-10.522 to -5.047], Standard Error of Mean 1.305
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Treatment contrast in LS mean (change), Adults; Test type: Superiority; p = 0.7768, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS mean = 0.710, 95% CI 2-sided [-1.118 to 2.538], Standard Error of Mean 0.933

2. Primary Outcome: Mean Change From Baseline in UAS7 at Week 12 (Observed Data) of Adolescent Subjects (FAS)
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized adolescent subjects who received at least one dose of study drug. Subjects were analyzed according to the treatment to which they were assigned at randomization. FAS was used for all efficacy variables, unless otherwise stated.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 2
Score | -17.39 (13.070) | -14.64 (14.662) | -13.84 (15.343) | -12.75 (18.738)

3. Secondary Outcome: Number and Proportion of Subjects With UAS7=0 Response at Week 12 (Multiple Imputation - Adults, Observed Data for Adolescents)
Description: The Urticaria Activity Score (UAS) is the sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. Complete UAS7 response is defined as UAS7 = 0.
  No Statistical analysis was planned for adolescent group.
Time Frame: Week 12
Population: FAS: Adults + Adolescents (observed data) = Total
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 315 | 322 | 318 | 108
Participants
  Adults: number analyzed (Participants) | 306 | 312 | 306 | 106
  Adults | 102 | 104 | 116 | 8
  Adolescents: number analyzed (Participants) | 9 | 10 | 12 | 2
  Adolescents | 3 | 3 | 0 | 1
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 5.680, 95% CI 2-sided [2.667 to 12.095]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.8430, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 0.840, 95% CI 2-sided [0.598 to 1.180]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 5.734, 95% CI 2-sided [2.694 to 12.207]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.8312, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio, log = 0.848, 95% CI 2-sided [0.605 to 1.188]

4. Secondary Outcome: Mean Change From Baseline in ISS7 at Week 12 (Multiple Imputation) of Adult Subjects (FAS)
Description: Improvement of severity of itch assessed as absolute change from baseline in ISS7 score at Week 12
  Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate)
  Negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: FAS: Adults
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 306 | 312 | 306 | 106
score | -8.502 (0.305) | -8.532 (0.301) | -8.921 (0.302) | -5.402 (0.514)
Statistical Analysis 1: Comparison: Ligelizumab 120 mg vs Placebo; Adults; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -3.100, 95% CI 2-sided [-4.271 to -1.929], Standard Error of Mean 0.597
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults; Test type: Superiority; p = 0.8366, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = 0.419, 95% CI 2-sided [-0.419 to 1.258], Standard Error of Mean 0.428
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Superiority — Adults; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -3.130, 95% CI 2-sided [-4.295 to -1.966], Standard Error of Mean 0.594
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults; Test type: Superiority; p = 0.8201, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = 0.389, 95% CI 2-sided [-0.444 to 1.222], Standard Error of Mean 0.425

5. Secondary Outcome: Mean Change From Baseline in ISS7 at Week 12 (Observed Data) of Adolescent Subjects, (FAS)
Description: Improvement of severity of itch assessed as absolute change from baseline in ISS7 score at Week 12
  Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate)
  Negative change from baseline indicates improvement.. No Statistical Analysis was planned for adolescent population.
Time Frame: Baseline, Week 12
Population: FAS: Adolescents
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 2
score | -8.40 (6.779) | -6.82 (7.404) | -5.10 (7.153) | -7.00 (9.899)

6. Secondary Outcome: Number and Proportion of Participants With DLQI Score of 0 - 1 at Week 12 (Multiple Imputation - Adults, Observed Data for Adolescents)
Description: Assessed as percentage of subjects achieving DLQI = 0-1, meaning, no impact on subjects quality of life at Week 12
  The Dermatology life Quality Index (DLQI) score range is 0 to 30, with 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
  No statistical anaylsis was planned for adolescent group.
Time Frame: Baseline, Week 12
Population: FAS: Adults + Adolescents (observed) = Total
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 315 | 323 | 318 | 109
Participants
  Adults: number analyzed (Participants) | 306 | 312 | 306 | 106
  Adults | 133 | 150 | 147 | 22
  Adolescents: number analyzed (Participants) | 9 | 11 | 12 | 3
  Adolescents | 3 | 6 | 2 | 1
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 2.747, 95% CI 2-sided [1.621 to 4.656]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.8586, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 0.836, 95% CI 2-sided [0.603 to 1.159]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 3.261, 95% CI 2-sided [1.929 to 5.513]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.5190, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 0.992, 95% CI 2-sided [0.717 to 1.373]

7. Secondary Outcome: Cumulative Number of Weeks of AAS7=0 up to Week 12 (Multiple Imputation) of Adult Subjects (FAS)
Description: Cumulative number of weeks that subjects achieve AAS7 = 0 responses between baseline and Week 12
  Angioedema Activity Score (AAS7) is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-15 (mean day sum score) where higher scores indicate increased angioedema activity.
Time Frame: Baseline, Week 12
Population: FAS: Adults
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 306 | 312 | 306 | 106
Weeks | 8.568 (0.235) | 8.912 (0.239) | 8.790 (0.239) | 6.475 (0.327)
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults; Test type: Superiority; p < .0001, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.323, 95% CI 2-sided [1.183 to 1.480]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults; Test type: Superiority; p = 0.7469, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 0.975, 95% CI 2-sided [0.904 to 1.051]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults; Test type: Superiority; p < .0001, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.376, 95% CI 2-sided [1.230 to 1.540]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults; Test type: Superiority; p = 0.3586, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.014, 95% CI 2-sided [0.941 to 1.092]

8. Secondary Outcome: Cumulative Number of Weeks of AAS7=0 up to Week 12 (Observed Data) of Adolescent Subjects (FAS)
Description: Cumulative number of weeks that subjects achieve AAS7 = 0 responses between baseline and Week 12
  Angioedema Activity Score (AAS7) is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-15 (mean day sum score) where higher scores indicate increased angioedema activity.
  No Statistical Analysis was planned.
Time Frame: Baseline, Week 12
Population: FAS: Adolescents
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 6 | 8 | 10 | 1
Weeks | 6.0 (4.94) | 7.3 (5.44) | 9.0 (3.50) | 11.0 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) monitoring was continued for at least 30 days following the last dose of study treatment or end of study visit (64 weeks), whichever is longer.
Description: An AE is any untoward medical occurrence, unfavorable, or unintended sign (including an abnormal laboratory finding), symptom, disease, or injury, temporally associated with the use of a marketed or investigational medicinal product, gene therapy, theragnostic product, or medical device, in patients, clinical-trial subjects, device users, or other persons, whether or not it is considered to be related to or due to the product.
Groups:
- QGE031 72mg: QGE031 72mg
- QGE031 120mg: QGE031 120mg
- Omalizumab 300mg: Omalizumab 300mg
- Placebo Only: Placebo only
- Transitioned to QGE031 120mg: Transitioned to QGE031 120mg
Arm/Group | QGE031 72mg | QGE031 120mg | Omalizumab 300mg | Placebo Only | Transitioned to QGE031 120mg
All-Cause Mortality (participants affected / at risk) | 0/316 | 0/324 | 0/319 | 0/109 | 0/102
Serious Adverse Events (participants affected / at risk) | 22/316 | 32/324 | 23/319 | 3/109 | 4/102
Other Adverse Events (participants affected / at risk) | 178/316 | 182/324 | 206/319 | 38/109 | 43/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 72mg (N=316) | QGE031 120mg (N=324) | Omalizumab 300mg (N=319) | Placebo Only (N=109) | Transitioned to QGE031 120mg (N=102)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 2 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 3 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 72mg (N=316) | QGE031 120mg (N=324) | Omalizumab 300mg (N=319) | Placebo Only (N=109) | Transitioned to QGE031 120mg (N=102)
Abdominal pain (Gastrointestinal disorders) | 1 | 6 | 9 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5 | 8 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 18 | 4 | 3
Nausea (Gastrointestinal disorders) | 8 | 9 | 10 | 1 | 2
Toothache (Gastrointestinal disorders) | 4 | 9 | 5 | 1 | 3
Vomiting (Gastrointestinal disorders) | 4 | 2 | 2 | 0 | 3
Fatigue (General disorders) | 4 | 6 | 8 | 0 | 1
Injection site erythema (General disorders) | 8 | 14 | 5 | 0 | 2
Injection site pain (General disorders) | 12 | 10 | 4 | 0 | 2
Injection site reaction (General disorders) | 15 | 15 | 7 | 0 | 6
Injection site swelling (General disorders) | 7 | 8 | 3 | 0 | 1
Pyrexia (General disorders) | 13 | 11 | 12 | 4 | 1
Bronchitis (Infections and infestations) | 6 | 3 | 7 | 1 | 1
COVID-19 (Infections and infestations) | 9 | 5 | 12 | 1 | 1
Gastroenteritis (Infections and infestations) | 9 | 5 | 6 | 3 | 2
Influenza (Infections and infestations) | 6 | 7 | 11 | 1 | 2
Nasopharyngitis (Infections and infestations) | 35 | 32 | 38 | 10 | 8
Rhinitis (Infections and infestations) | 1 | 1 | 7 | 0 | 2
Sinusitis (Infections and infestations) | 6 | 8 | 6 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 20 | 24 | 28 | 4 | 1
Urinary tract infection (Infections and infestations) | 11 | 10 | 12 | 3 | 5
Contusion (Injury, poisoning and procedural complications) | 7 | 1 | 4 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 7 | 0 | 1
Alanine aminotransferase increased (Investigations) | 8 | 10 | 5 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 8 | 4 | 0 | 1
Blood creatinine increased (Investigations) | 6 | 8 | 11 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 7 | 4 | 0 | 2
SARS-CoV-2 test negative (Investigations) | 2 | 7 | 7 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 5 | 5 | 8 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 19 | 16 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 9 | 16 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7 | 3 | 0
Dizziness (Nervous system disorders) | 12 | 8 | 2 | 2 | 1
Headache (Nervous system disorders) | 40 | 30 | 39 | 6 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 8 | 6 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 14 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 18 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 8 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 4 | 9 | 7 | 2 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 4 | 6 | 12 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 4 | 9 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 6 | 8 | 11 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 17 | 15 | 10 | 2 | 3
Hypertension (Vascular disorders) | 5 | 6 | 8 | 2 | 1

LIMITATIONS AND CAVEATS:
The difference of 4 subjects between RAN (1034) vs FAS (1030) is due to mis-randomization of 4 subjects. These subjects did not receive Ligelizumab and hence rightfully not included in FAS (though included in RAN).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT03580369/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03580369/SAP_001.pdf